CLINICAL TRIAL: NCT01546935
Title: SEA022 Oseltamivir Treatment in Children Under One Year of Age With Moderate or Severe Influenza Lower Respiratory Tract Infection - a Clinical and Pharmacokinetic Study.
Brief Title: Oseltamivir for Influenza Lower Respiratory Tract Infection in Children Under One
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Study drugs (Oseltamivir suspension from Roche) were unavailable
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SEA022
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Influenza
Keywords: Influenza; Oseltamivir; Lower tract respiratory infection
MeSH Terms: conditions — Influenza, Human | interventions — Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oseltamivir (Experimental): The dose of Oseltamivir will be 3 mg/kg 12 hourly for 5 days (seasonal influenza and 2009 H1N1) or 10 days (avian influenza) for children whose renal function is ≥ 30 mls/min/1.73m2.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Oseltamivir — The dose of Oseltamivir will be 3 mg/kg 12 hourly for 5 days (seasonal influenza and 2009 H1N1) or 10 days (avian influenza) for children whose renal function is ≥ 30 mls/min/1.73m2.
  Other Names: Tamiflu

SUMMARY:
Currently, there is no treatment for children less than one year of age with influenza related lower respiratory tract infection that is either considered standard or registered in any country. This dismal scenario exists even though influenza related LRTI is a significant illness causing morbidity and mortality, especially in children less than 6 months of age. Avian influenza has been reported rarely in children less than one.

There are no data in Vietnam and very few data in Thailand on the burden of influenza in children less than one. This young age group suffers high mortality. Oseltamivir may be beneficial in such children. This is basis of this trial.

DETAILED DESCRIPTION:
There are limited data from Thailand on the aetiology of LRTI but no data on mortality of hospitalised children. Thai children < 1 year accounted for circa one third of LRTIs in children who were treated as out or inpatients in whom influenza was isolated in 6 (2.7%) of 271 children and RSV in 44 (20%). At the Queen Sirikit hospital, Bangkok, influenza A and B and RSV accounted for approximately 11% (9/80), 2.5% (2/80) and 6% (5/80) of children < 1 year, respectively. This study included children with underlying diseases like congenital heart disease and chronic lung disease. A small laboratory series of 110 children at Siriraj hospital with LRTIs infections (Pilaipan Puthavathana, personal communication) identified RSV A/B (17%), metapneumovirus (14%), parainfluenza 1 (12%) and adenovirus (12%), influenza B (6%), influenza A (4%), coronaviruses (3%), Parainfluenza 3 (2%) and 2 (0%).

The number of drugs registered for treating influenza is limited to oral Oseltamivir, amantadine and rimantadine and inhaled zanamivir. As a result of the 2009 influenza A/H1N1, clinical guidelines have been updated to include children less than one years old . However, regulatory studies of oseltamivir excluded children under 1 year based on preclinical data in rats in which there were deaths in young rats (7 days old) but none in 14 days old rats given large doses of Oseltamivir. Higher concentrations of Oseltamivir were found in the brains of the younger rats which was thought to be due immaturity of the blood brain barrier.

There is, however, some clinical experience with Oseltamivir in the under ones from Japan, Thailand, Germany , the USA , and additional experience with 2009 pH1N1 . The doses used were 2 mg/kg bid which is consistent with the dose recommended in the UK for children who weigh less than 15 kg (30 mg bid for 5 days). At the Queen Sirikit hospital, Oseltamivir has been given to a very small number of children < 1 year with severe influenza with good effect (T. Chotpitayasunondh, unpublished observations). This experience is similar to that of others i.e. good clinical outcomes and apparently good tolerability.

An Oseltamivir pharmacokinetic study in children age 1-5 years showed that the dose of 2 mg/kg resulted in plasma-concentration time curves (AUC) similar to the AUC accepted in adult. However, the younger the child, the lower the AUC level; never the less, there are still insufficient pharmacokinetics data in children under one year .

The clinical significance of reduced in vitro sensitivity is unclear owing to the paucity of human data but these mutations are likely to result in reduced antiviral efficacy of Oseltamivir and the adamantanes against H1N1. Furthermore, amantadine treatment of influenza frequently results in the rapid development of amantadine resistance in both H1N1 and H2N3 viruses, resulting in continued virus replication, thus, making this drug less than ideal for treating influenza. Currently, there is limited adamantane resistant H1N1 but widespread adamantane resistant in H3N2. H3N2 and influenza B remain sensitive to Oseltamivir. The adamantanes have no activity against influenza B.

The emergence of resistance poses difficulties for the treatment of influenza in children less than one but oseltamivir represents at present the optimal choice for treating such children. Therefore, this protocol will assess the effect of oral Oseltamivir at doses recommended by the WHO to see if they are applicable to Thai children.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by a parent/legal guardian.
* Children less than 12 months of age when first seen with a LRTI of moderate or severe severity and virologically proven influenza on a respiratory specimen.
* History of fever within 14 days prior to presentation (note: a fever at presentation is not required) plus any two of the following:
* Cough
* Difficulty breathing / shortness of breath
* Increased respiratory rate for that age:
* > 60/min, age < 2 months
* > 50/min, age 2 - < 12 months,
* Intercostal recession
* Use of accessory muscles
* Nasal flare/grunting
* Crepitations with or without wheezing
* A consistent abnormal chest X ray e.g. new infiltrate, hyperinflation

Virological evidence of influenza on the following test:

* A positive commercial rapid test confirmed twice for influenza on respiratory specimens from 2 different anatomical sites*

  * Any one of the following constitutes an acceptable respiratory specimen:
* NPA
* NP swab
* throat swab
* endotracheal aspirate
* bronchoalveolar lavage sample

Exclusion Criteria:

Exclusion criteria for children with non avian influenza

These are:

* Known allergy to Oseltamivir
* Age ≥ 12 months on the day of hospital admission
* Illness duration > 14 days on the day of hospital admission
* Creatinine clearance < 10 mls/min/1.73m2, including a requirement for dialysis or haemofiltration Exclusion criteria for children with avian influenza

These are:

* Known allergy to Oseltamivir
* Age ≥ 12 months on the day of hospital admission
* Informed consent not obtained

Patients with the following can be enrolled:

* underlying illnesses
* if prescribed Oseltamivir prior to presentation
* for avian influenza only: creatinine clearance < 10 mls/min/1.73m2, including a requirement for dialysis or haemofiltration

Max Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Viral clearance | 5-10 days
  * Viral clearance on Day 5 (human influenza) on a throat swab, assessed by RT PCR.
  * Viral clearance on Day 10 (avian influenza) on a throat swab, assessed by RT PCR.
Pharmacokinetics of Oseltamivir | Day 0 and Day 9
  • Cmax, Tmax, AUC, apparent volume of distribution, clearance, terminal elimination half-life

SECONDARY OUTCOMES:
Viral end points | 5-10 days
  * Time to viral clearance on a throat swab, assessed by RT PCR.
  * The time to no detectable influenza virus by culture for the throat swab.
  * Change in viral load (log10 copies/mL) over time for all virological samples (lower limit of detection: 1000 copies/mL)
  * Viral susceptibility of cultured influenza virus to antiviral drugs at baseline and post treatment, assessed by genotypical and phenotypical analyses
Clinical Efficacy Endpoints | 5-10 days
  * Time to fever clearance
  * In hospital mortality and mortality by follow up
  * Time to death
  * Time to trans cutaneous O2 saturation of ≥ 95% on room air
  * Clinical course: pneumothorax, encephalitis/encephalopathy
  * Number of days in hospital
  * Number of days ventilated
Safety Endpoints | 5-10 days
  * Documented serious adverse events (SAEs) and relationships to oseltamivir
  * AEs leading to drug withdrawal
  * Grade 3 & 4 clinical and laboratory AEs that are probably or definitely related to oseltamivir
  * Skin rashes of any grade
  * Changes in haematological and biochemical parameters over time

CONTACTS AND LOCATIONS:
Overall Officials: Kulkanya Chokephaibulkit, MD, Principal Investigator — Siriraj Hospital; Piyarat Suntarattiwong, MD, Principal Investigator — Queen Sirikit National Institute of Health
Locations (2):
- Thailand (2):
  - Queen Sirikit National Institute of Child Health, Bangkok, Bangkok
  - Faculty of Medicine Siriraj Hospital, Bangkok, Bangkok